CLINICAL TRIAL: NCT06376552
Title: The Use of Artificial Intelligence for the Prioritization of Causative Genetic Background in a Brugada Syndrome Cohort: an Observational Retrospective Study
Brief Title: Artificial Intelligence for the Prioritization of Genetic Background in Brugada Syndrome
Acronym: AI4Cardio
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Chiara Di Resta, PhD, IRCCS San Raffaele
Other Study IDs: AI4Cardio
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Brugada Syndrome
MeSH Terms: conditions — Brugada Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BrS Patients: The 200 BS patients have been selected and clinically evaluated by Department of Cardiac Electrophysiology and Arrhythmology, San Raffaele Hospital, for the presence of a type I electrocardiogram (ECG), either spontaneous or induced by flecainide or ajmaline. Morphologic and functional characteristics of the heart have been analysed in all patients by trans-thoracic echocardiography and stress test to rule out patients with Arrhythmogenic Right Ventricular Dysplasia and ischemic heart disease. Among clinical characteristics, 12-lead signal averaged ECG parameters and all possible risk factors have been evaluated. Electrophysiological study has been performed in spontaneous BS pattern 1 ECG patients or patients with induced BS pattern 1 ECG and at least one risk factor. In patients with higher susceptibility for the induced Ventricular Tachycardia, ICD has been implanted.

SUMMARY:
Brugada Syndrome (BS) is an inherited heart condition that can cause sudden cardiac arrest in young individuals. It's diagnosed through specific changes seen on an electrocardiogram (ECG). Currently, the only treatment option is a cardioverter defibrillator (ICD). Despite advances, much about BS remains unclear, including its genetic basis. This study aims to use advanced genetic sequencing and artificial intelligence to uncover new genetic factors contributing to BS. By understanding these factors better, we hope to improve risk assessment and treatment for affected individuals.

DETAILED DESCRIPTION:
Brugada Syndrome (BS) is an inherited cardiac electrical disorder that can cause syncope and sudden cardiac arrest in young asymptomatic individuals. It is suspected to contribute to 4-12% of cases of sudden cardiac death in the general population. Diagnosis relies on identifying a type I ECG pattern characterized by ST-segment elevation with a coved morphology in the right precordial leads. The prevalence in Western countries is estimated at 1:5000. Currently, implantation of a cardioverter defibrillator (ICD) is the only treatment option, but risk stratification guidelines remain incomplete, particularly for asymptomatic individuals.

BS is inherited as an autosomal dominant trait with incomplete penetrance. While 23 genes have been associated with BS susceptibility, 70% of patients remain genetically uncharacterized, suggesting a more complex inheritance pattern. Genetics have not been incorporated into risk stratification guidelines, despite evidence linking certain genetic variants to higher arrhythmic risk. This knowledge gap underscores the importance of expanding our understanding of BS genetics to enhance diagnostic sensitivity and patient management.

This protocol builds upon preliminary data from a study granted by the Italian Ministry of Health (GR-2016-02362316), in which next-generation sequencing (NGS) was used to investigate the entire coding regions (Whole Exome Sequencing_WES) of 200 BS patients. The study aimed to identify new BS candidate genes and characterize the genetic basis of the condition.

The cohort was selected based on the presence of a type I ECG, confirmed either spontaneously or induced by flecainide or ajmaline. Patients underwent thorough cardiac evaluations to rule out other conditions. Follow-up included yearly assessments and more frequent evaluations for patients with a higher risk of ventricular tachycardia.

A large number of genetic variants were identified by exploiting WES, prompting the use of Artificial Intelligence (AI) to prioritize the sequencing data. AI techniques, including advanced algorithms and machine learning, can streamline the identification of potentially disease-causing genetic variations by filtering out common variants, predicting pathogenicity, and integrating clinical data.

Given that over 70% of BS patients remain genetically undiagnosed, high-throughput sequencing approaches are crucial for a comprehensive understanding of BS genetics. This study aims to contribute to the identification of new genetic factors and improve risk stratification for affected patients. All sequencing data for this project have been generated and will be analyzed using AI, with no further patients to be enrolled or sequenced.

ELIGIBILITY:
Inclusion Criteria:

* The 200 BS patients have been selected and clinically evaluated based on the presence of a type I electrocardiogram (ECG), either spontaneous or induced by flecainide or ajmaline.

Exclusion Criteria:

* No exclusion criteria are adopted for this study. The entire previously sequenced cohort of 200 BS patients will be investigated and considered, exploiting AI approach for the prioritization of the sequencing available data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 BS patients.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-06-06 (Actual)

PRIMARY OUTCOMES:
New candidate genes, likely associated with Brugada Syndrome using an AI based approach. | 1 year
  Prioritization of genetic variations underlying the BS phenotype: the whole exome data of 200 BS previously sequenced will be prioritized using an AI- based approach, developed by the collaborators in UniMIB.

SECONDARY OUTCOMES:
Identification of genetic risk factors associated with the worse phenotype. | 1 year
  Correlation of the new putative genes and the clinical variables, previously collected in a comprehensive database for this study.

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Di Resta, PhD, Principal Investigator — IRCCS San Raffaele Hospital
Locations (2):
- Italy (2):
  - IRCCS San Raffaele, Milan
  - Milano-Bicocca University, Milan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Di Resta C, Pietrelli A, Sala S, Della Bella P, De Bellis G, Ferrari M, Bordoni R, Benedetti S. High-throughput genetic characterization of a cohort of Brugada syndrome patients. Hum Mol Genet. 2015 Oct 15;24(20):5828-35. doi: 10.1093/hmg/ddv302. Epub 2015 Jul 28. PMID 26220970
- [Background] Sommariva E, Pappone C, Martinelli Boneschi F, Di Resta C, Rosaria Carbone M, Salvi E, Vergara P, Sala S, Cusi D, Ferrari M, Benedetti S. Genetics can contribute to the prognosis of Brugada syndrome: a pilot model for risk stratification. Eur J Hum Genet. 2013 Sep;21(9):911-7. doi: 10.1038/ejhg.2012.289. Epub 2013 Jan 16. PMID 23321620
- [Background] Di Resta C, Berg J, Villatore A, Maia M, Pili G, Fioravanti F, Tomaiuolo R, Sala S, Benedetti S, Peretto G. Concealed Substrates in Brugada Syndrome: Isolated Channelopathy or Associated Cardiomyopathy? Genes (Basel). 2022 Sep 28;13(10):1755. doi: 10.3390/genes13101755. PMID 36292641